CLINICAL TRIAL: NCT00299182
Title: Phase 1/2 Study of AMG 531 to Evaluate the Safety, Efficacy, and Pharmacokinetics in Patients With Aggressive Non-Hodgkin's Lymphoma Receiving R-HyperCVAD Alternating With R-Ara-C/MTX
Brief Title: Study of AMG 531 to Evaluate the Safety & Efficacy in Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005-0146
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Results first posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-08

CONDITIONS: Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Lymphoma; Mantle Cell Lymphoma; AMG 531; Romiplostim; Placebo; R-HyperCVAD; R-Ara-C/MTX; Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Methotrexate; Rituximab; Vincristine; Decadron; Neosar; AD; Hydroxydaunomycin hydrocholoride; Ara-C; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell | interventions — romiplostim; Rituximab; Cyclophosphamide; Vincristine; Doxorubicin; Dexamethasone; Calcium Dobesilate; Methotrexate; Cytarabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 mcg/ kg AMG531 Pre & Post Chemotherapy (Experimental): Cycle 1, Chemotherapy (R-HyperCVAD) alone.
  Cycle 2, Chemotherapy (R-Ara-C/MTX), followed by 1 mcg/ kg AMG 531 subcutaneously on days -5 and 5 (Arm A)
  R-HyperCVAD alternating with R-Ara-C/MTX where R-HyperCVAD is Rituximab 375 mg/m^2; plus Cyclophosphamide 300 mg/m^2, Vincristine 1.4 mg/m^2, Doxorubicin (Adriamycin) 50 mg/m^2, and Dexamethasone 40 mg (CVAD), Mesna 600mg/m^2; and, R-Ara-C/MTX is Rituximab 375 mg/m^2, Cytarabine 3 g/m^2 and Methotrexate 200 mg/m^2.
  Interventions: Drug: AMG 531; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Dexamethasone; Drug: Methotrexate; Drug: Cytarabine
- 3 mcg/ kg AMG531 Pre & Post Chemotherapy (Experimental): Cycle 1, Chemotherapy (R-HyperCVAD) alone.
  Cycle 2, Chemotherapy (R-Ara-C/MTX), followed by 3 mcg/ kg AMG 531 subcutaneously on days -5 and 5 (Arm A)
  R-HyperCVAD alternating with R-Ara-C/MTX where R-HyperCVAD is Rituximab 375 mg/m^2; plus Cyclophosphamide 300 mg/m^2, Vincristine 1.4 mg/m^2, Doxorubicin (Adriamycin) 50 mg/m^2, and Dexamethasone 40 mg (CVAD), Mesna 600mg/m^2; and, R-Ara-C/MTX is Rituximab 375 mg/m^2, Cytarabine 3 g/m^2 and Methotrexate 200 mg/m^2.
  Interventions: Drug: AMG 531; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Dexamethasone; Drug: Methotrexate; Drug: Cytarabine
- 10 mcg/ kg AMG531 Pre & Post Chemotherapy (Experimental): Cycle 1, Chemotherapy (R-HyperCVAD) alone.
  Cycle 2, Chemotherapy (R-Ara-C/MTX), followed by 10 mcg/ kg AMG 531 subcutaneously on days -5 and 5 (Arm A)
  R-HyperCVAD alternating with R-Ara-C/MTX where R-HyperCVAD is Rituximab 375 mg/m^2; plus Cyclophosphamide 300 mg/m^2, Vincristine 1.4 mg/m^2, Doxorubicin (Adriamycin) 50 mg/m^2, and Dexamethasone 40 mg (CVAD), Mesna 600mg/m^2; and, R-Ara-C/MTX is Rituximab 375 mg/m^2, Cytarabine 3 g/m^2 and Methotrexate 200 mg/m^2.
  Interventions: Drug: AMG 531; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Dexamethasone; Drug: Methotrexate; Drug: Cytarabine
- Placebo (Arm A & Arm B) with Chemotherapy (Placebo Comparator): Placebo Pre and Post (Arm A), or Post (Arm B) Chemotherapy
  Cycle 1, Chemotherapy (R-HyperCVAD) alone.
  Cycle 2, Chemotherapy (R-Ara-C/MTX), followed by placebo subcutaneously on days -5 and 5 (Arm A) or days 5 and 7 (Arm B)
  R-HyperCVAD alternating with R-Ara-C/MTX where R-HyperCVAD is Rituximab 375 mg/m^2; plus Cyclophosphamide 300 mg/m^2, Vincristine 1.4 mg/m^2, Doxorubicin (Adriamycin) 50 mg/m^2, and Dexamethasone 40 mg (CVAD), Mesna 600mg/m^2; and, R-Ara-C/MTX is Rituximab 375 mg/m^2, Cytarabine 3 g/m^2 and Methotrexate 200 mg/m^2.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Dexamethasone; Drug: Methotrexate; Drug: Cytarabine; Drug: Placebo
- 1 mcg/ kg AMG531 Post Chemotherapy (Experimental): Cycle 1, Chemotherapy (R-HyperCVAD) alone.
  Cycle 2, Chemotherapy (R-Ara-C/MTX), followed by 1 mcg/ kg AMG 531 subcutaneously on days 5 and 7 (Arm B)
  R-HyperCVAD alternating with R-Ara-C/MTX where R-HyperCVAD is Rituximab 375 mg/m^2; plus Cyclophosphamide 300 mg/m^2, Vincristine 1.4 mg/m^2, Doxorubicin (Adriamycin) 50 mg/m^2, and Dexamethasone 40 mg (CVAD), Mesna 600mg/m^2; and, R-Ara-C/MTX is Rituximab 375 mg/m^2, Cytarabine 3 g/m^2 and Methotrexate 200 mg/m^2.
  Interventions: Drug: AMG 531; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Dexamethasone; Drug: Methotrexate; Drug: Cytarabine
- 3 mcg/ kg AMG531 Post Chemotherapy (Experimental): Cycle 1, Chemotherapy (R-HyperCVAD) alone.
  Cycle 2, Chemotherapy (R-Ara-C/MTX), followed by 3 mcg/ kg AMG 531 subcutaneously on days 5 and 7 (Arm B)
  R-HyperCVAD alternating with R-Ara-C/MTX where R-HyperCVAD is Rituximab 375 mg/m^2; plus Cyclophosphamide 300 mg/m^2, Vincristine 1.4 mg/m^2, Doxorubicin (Adriamycin) 50 mg/m^2, and Dexamethasone 40 mg (CVAD), Mesna 600mg/m^2; and, R-Ara-C/MTX is Rituximab 375 mg/m^2, Cytarabine 3 g/m^2 and Methotrexate 200 mg/m^2.
  Interventions: Drug: AMG 531; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Dexamethasone; Drug: Methotrexate; Drug: Cytarabine
- 10 mcg/ kg AMG531 Post Chemotherapy (Experimental): Cycle 1, Chemotherapy (R-HyperCVAD) alone.
  Cycle 2, Chemotherapy (R-Ara-C/MTX), followed by 10 mcg/ kg AMG 531 subcutaneously on days 5 and 7 (Arm B)
  R-HyperCVAD alternating with R-Ara-C/MTX where R-HyperCVAD is Rituximab 375 mg/m^2; plus Cyclophosphamide 300 mg/m^2, Vincristine 1.4 mg/m^2, Doxorubicin (Adriamycin) 50 mg/m^2, and Dexamethasone 40 mg (CVAD), Mesna 600mg/m^2; and, R-Ara-C/MTX is Rituximab 375 mg/m^2, Cytarabine 3 g/m^2 and Methotrexate 200 mg/m^2.
  Interventions: Drug: AMG 531; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Dexamethasone; Drug: Methotrexate; Drug: Cytarabine

INTERVENTIONS:
Drug: AMG 531 — Arm A: AMG531 - 1, 3, or 10 mcg/kg subcutaneous injection administered on on days -5 and 5 (pre and post chemotherapy dose) beginning with Cycle 2; OR, Arm A: AMG531 - 1, 3, or 10 mcg/kg subcutaneous injection administered on on days 5 and 7 (post chemotherapy doses only) beginning with Cycle 2.
  Other Names: Romiplostim
  Arms: 1 mcg/ kg AMG531 Post Chemotherapy; 1 mcg/ kg AMG531 Pre & Post Chemotherapy; 10 mcg/ kg AMG531 Post Chemotherapy; 10 mcg/ kg AMG531 Pre & Post Chemotherapy; 3 mcg/ kg AMG531 Post Chemotherapy; 3 mcg/ kg AMG531 Pre & Post Chemotherapy
Drug: Rituximab — 375 mg/m^2 by vein over 4-6 hour infusion day 1, each cycle.
  Other Names: Rituxan
Drug: Cyclophosphamide — 300 mg/m^2 by vein over 3 hours every 12 hours for 6 doses (days 2-4), Cycles 1,3, & 5.
  Other Names: Cytoxan; Neosar
Drug: Vincristine — 1.4 mg/m^2/dose (maximum 2 mg) by vein over 15 minutes Days 5 and 12, Cycles 1,3,& 5.
Drug: Doxorubicin — 50 mg/m^2/dose by vein over 15 minutes on Day 5 or by continuous infusion over 24-48 hours (days 5-6), Cycles 1,3,& 5.
  Other Names: AD; Hydroxydaunomycin hydrocholoride
Drug: Dexamethasone — 40 mg/day by mouth or by vein days 2-5 and 12-15, Cycles 1,3,& 5.
  Other Names: Decadron
Drug: Methotrexate — 200 mg/m^2 by vein over 2 hours followed by 800 mg/m^2 over 22 hours Day 2, Cycles 2, 4 & 6.
Drug: Cytarabine — 3 g/m^2 by vein over 2 hours every 12 hours for 4 doses, days 3 & 4; OR,1 g/m^2 by vein over 2 hours every 12 hours for 4 doses, days 3 & 4 for patients > 60 years and for patients with serum creatinine > 1.5 mg/dL; Cycles 2,4,& 6.
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride
Drug: Placebo — Arm A: Placebo - subcutaneous injection administered on days -5 and 5 (pre and post chemotherapy dose) beginning with Cycle 2; OR, Arm B: Placebo - subcutaneous injection administered on days 5 and 7 (post chemotherapy doses only) beginning with Cycle 2.
  Arms: Placebo (Arm A & Arm B) with Chemotherapy

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of AMG 531 that can be given to treat thrombocytopenia (low platelet counts) in patients who have received chemotherapy. Researchers will also look at the safety and effectiveness of AMG 531.

Primary Objectives:

1. To determine the clinical safety and tolerability of AMG 531 administered following chemotherapy (R-HyperCVAD alternating with R-Ara-C/MTX) in patients with non-Hodgkin's lymphoma.
2. To determine an optimal biologic dose (OBD) of AMG 531 in patients receiving R-HyperCVAD and R-Ara-C/MTX.
3. To evaluate the effects of AMG 531 on the degree and duration of thrombocytopenia and platelet recovery following chemotherapy(chemo).

Secondary Objectives:

1. To evaluate limited pharmacokinetics of AMG 531 administered by S.C. route with chemotherapy.

DETAILED DESCRIPTION:
Platelets are cells that help make the blood clot. A decrease in platelets can cause bleeding, which may prevent or delay a patient from receiving chemotherapy. R-HyperCVAD (rituximab, cyclophosphamide, vincristine, doxorubicin, and dexamethasone) and R-Ara-C/MTX (rituximab, cytarabine, and methotrexate) are two chemotherapy regimens that are known to increase the risk of lower platelet counts. Researchers want to find out if AMG 531 can lower the risk and severity of this side effect. AMG 531 is a protein that stimulates platelet production.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete medical history and physical exam, including measurement of vital signs (temperature, pulse, breathing rate, and blood pressure). You will have blood collected (about 3 teaspoons) for routine tests. Radiologic tests such as CT or MRI scans will be done as needed. Women who are able to have children must have a negative blood pregnancy test.

You will also have about 1 teaspoon of blood drawn to see if the you have antibodies to the study drug.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of four treatment groups. These 4 groups will also be split into 2 separate subgroups (Arm A and Arm B). Participants in Arm A will either receive AMG 531 or placebo on Day -5 (5 days before chemotherapy starts) and Day 5 (5 days after chemotherapy starts). A placebo is a substance that looks like the study drug but which has no active ingredients. Every 2 out of 3 participants in Arm A will receive AMG 531. One out of every 3 participants in Arm A will receive placebo.

Participants in Arm B will receive either AMG 531 or placebo on Day 5 and 7. Every 2 out of 3 participants in Arm B will receive AMG 531. One out of every 3 participants in Arm B will receive placebo. The dose of AMG 531 that participants in both Arms A and B receive will depend on when they enroll on the study. There are 3 different dose levels of AMG 531 being studied. Each new group of participants will receive a higher dose than the previous group.

All participants will receive treatment with R-HyperCVAD and R-Ara-C/MTX chemotherapy by vein in alternating cycles. In Cycle 1, all participants will receive R-HyperCVAD by itself. Each cycle is 3 weeks long.

Three (3) weeks later, in Cycle 2, all participants will receive either AMG 531 or placebo following R-Ara-C/MTX. The AMG 531/placebo will be given as an injection under the skin on Days -5 and 5 (Arm A) or on Days 5 and 7 (Arm B). After 2 cycles of treatment, based on response of the disease and tolerance to the treatment, all participants may be able to receive up to 4 more cycles of chemotherapy followed by AMG 531. For Cycles 3-6, you will follow the same schedule of therapy as in the first 2 cycles. The dose of AMG 531 may be increased at one time point during the study based on the response of the platelet counts.

Blood (about 1 teaspoon) will be collected for the evaluation of anti-AMG 531 antibody status at the end of Cycles 2 and 4. You will be taken off the study if your disease gets worse or intolerable side effects occur. The number of blood tests drawn will depend on your clinical condition. These samples (about 1 teaspoon each) will be taken at least 2 times a week and as often as once a day during anticipated periods of low blood cell counts.

At the end of the study, you will have an interim medical history and physical exam, including measurement of vital signs. You will have blood (about 1 teaspoon) drawn for routine end-of-study analysis. Blood (about 1 teaspoon) will also be collected for the evaluation of anti-AMG 531 antibody status.

This is an investigational study. R-HyperCVAD and R-Ara-C/MTX are commercially available chemotherapy drugs. AMG 531 is not FDA approved or commercially available. At this time, AMG 531 is being used in this study for research purposes only. About 36 evaluable patients (maximum of 50 patients) will take part in this study. All will be enrolled at University of Texas (UT) M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of previously untreated aggressive non-Hodgkin's lymphoma, including patients with mantle cell lymphoma, who will be or are receiving treatment with R-HyperCVAD and R-Ara-C/MTX. Patients in whom Rituximab is not used, due to contraindication, will be eligible. Patients whose therapy was switched to (R)Hyper-CVAD after initial treatment with (R)CHOP, because of aggressive disease will also be eligible for the study.
2. Patients age >/= 18 years.
3. Karnofsky Performance Scale >/= 70.
4. Adequate hematologic (ANC >/= 1000/mm(3), platelet count >/= 100,000/mm(3) and Hgb >/= 8gm/dL), renal (serum creatinine < 2mg/dL), and hepatic functions (total bilirubin </= 2 times, serum glutamate pyruvate transaminase (SGPT) or serum glutamate oxaloacetate transaminase (SGOT) </= 3 times the upper limit of the respective normal range).
5. Patients (male and female) with childbearing potential (defined as not post-menopausal for 12 months or no previous surgical sterilization) must use adequate birth control.
6. Institutional Review Board (IRB)-approved signed informed consent.

Exclusion Criteria:

1. Pregnant or lactating women.
2. History of Central Nervous System (CNS) involvement.
3. Co-morbid medical or psychiatric illnesses that preclude treatment with intense dose chemotherapy.
4. Patients with history of deep vein thrombosis (DVT) or pulmonary embolus.
5. History of any platelet disorders including Idiopathic thrombocytopenic purpura (ITP), Thrombotic thrombocytopenic purpura (TTP) or bleeding disorders.
6. Prior surgery or Radiation Therapy (RT) within 2 weeks of study entry.
7. Patients with significant cardiac disease (New York Heart Association (NYHA) Class III or IV), dysrrhythmia, or recent history of myocardial ischemia (MI) or ischemia, transient ischemic attack or cerebrovascular accident (CVA) within the previous 6 months of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center official website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2, 2006 to February 1, 2010. All recruitment done at the University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: The protocol is designed to combine the placebo of Arm A and Arm B.
Period: Overall Study
Arm/Group | 1 mcg/ kg AMG531 Pre & Post Chemotherapy | 3 mcg/ kg AMG531 Pre & Post Chemotherapy | 10 mcg/ kg AMG531 Pre & Post Chemotherapy | Placebo (Arm A & Arm B) With Chemotherapy | 1 mcg/ kg AMG531 Post Chemotherapy | 3 mcg/ kg AMG531 Post Chemotherapy | 10 mcg/ kg AMG531 Post Chemotherapy
Started | 6 | 4 | 6 | 14 | 8 | 7 | 5
Completed | 6 | 4 | 4 | 14 | 5 | 4 | 4
Not Completed | 0 | 0 | 2 | 0 | 3 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 2 | 0
Not completed — Chemotherapy Changed | 0 | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Not Eligible | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of the 41 participants, 36 received treatment with the study drug as per protocol and were evaluable for response and toxicity; 5 participants received only one dose and were evaluable for toxicity only.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 mcg/ kg AMG531 Pre & Post Chemotherapy | 3 mcg/ kg AMG531 Pre & Post Chemotherapy | 10 mcg/ kg AMG531 Pre & Post Chemotherapy | Placebo (Arm A & Arm B) With Chemotherapy | 1 mcg/ kg AMG531 Post Chemotherapy | 3 mcg/ kg AMG531 Post Chemotherapy | 10 mcg/ kg AMG531 Post Chemotherapy | Total
Number analyzed (Participants) | 6 | 4 | 4 | 14 | 5 | 4 | 4 | 41
Age, Continuous [Median (Full Range); unit: years] | 57 [18 to 61] | 58 [40 to 73] | 59 [54 to 71] | 56 [28 to 73] | 51 [33 to 61] | 57 [18 to 67] | 56 [53 to 60] | 56 [18 to 73]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Between 18 and 65 years | 5 | 3 | 3 | 10 | 5 | 2 | 4 | 32
  >=65 years | 0 | 1 | 1 | 4 | 0 | 1 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3 | 4 | 0 | 1 | 11
  Male | 5 | 2 | 4 | 11 | 1 | 4 | 3 | 30
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 4 | 14 | 5 | 4 | 4 | 41

OUTCOME MEASURES:

1. Primary Outcome: Platelet (PLT) Nadir
Description: Blood counts were performed at least two times a week and when clinically indicated during the study and daily when PLT count is < 50K/μL until recovery (two consecutive counts showing upward trend). The optimal biologic dose was defined as the dose of AMG 531 at which the greatest proportion of patients avoided grade 4 thrombocytopenia (Platelet nadir < 25K/μL) in the absence of platelet transfusion in the blinded study cycle.
Time Frame: Prior to start of treatment and then at least 2 times a week during treatment until end of cycle 2 (1 cycle = 21 days)
Measure: Mean (Standard Error); unit: K/μL
Groups:
- Arm A 1mcg/kg; ARM A 3mcg/kg: Cycle 1, Chemotherapy (R-HyperCVAD) alone.
  Cycle 2, Chemotherapy (R-Ara-C/MTX), followed by either 1 mcg/kg or 3 mcg/kg or 10 mcg/kg AMG531 subcutaneously on days -5 and 5 (Arm A)
  R-HyperCVAD alternating with R-Ara-C/MTX where R-HyperCVAD is Rituximab 375 mg/m^2; plus Cyclophosphamide 300 mg/m^2, Vincristine 1.4 mg/m^2, Doxorubicin (Adriamycin) 50 mg/m^2, and Dexamethasone 40 mg (CVAD), Mesna 600mg/m^2; and, R-Ara-C/MTX is Rituximab 375 mg/m^2, Cytarabine 3 g/m^2 and Methotrexate 200 mg/m^2.
- Arm A 10mcg/kg; Arm B 1mcg/kg; Arm B 3mcg/kg; Arm B 10mcg/kg: Cycle 1, Chemotherapy (R-HyperCVAD) alone.
  Cycle 2, Chemotherapy (R-Ara-C/MTX), followed by either 1 mcg/kg or 3 mcg/kg or 10 mcg/kg AMG531 subcutaneously on days 5 and 7 (Arm B)
  R-HyperCVAD alternating with R-Ara-C/MTX where R-HyperCVAD is Rituximab 375 mg/m^2; plus Cyclophosphamide 300 mg/m^2, Vincristine 1.4 mg/m^2, Doxorubicin (Adriamycin) 50 mg/m^2, and Dexamethasone 40 mg (CVAD), Mesna 600mg/m^2; and, R-Ara-C/MTX is Rituximab 375 mg/m^2, Cytarabine 3 g/m^2 and Methotrexate 200 mg/m^2.
- Placebo: Placebo Pre and Post (Arm A), or Post (Arm B) Chemotherapy Cycle 1, Chemotherapy (R-HyperCVAD) alone. Cycle 2, Chemotherapy (R-Ara-C/MTX), followed by placebo subcutaneously on days -5 and 5 (Arm A) or days 5 and 7 (Arm B) R-HyperCVAD alternating with R-Ara-C/MTX where R-HyperCVAD is Rituximab 375 mg/m^2; plus Cyclophosphamide 300 mg/m^2, Vincristine 1.4 mg/m^2, Doxorubicin (Adriamycin) 50 mg/m^2, and Dexamethasone 40 mg (CVAD), Mesna 600mg/m^2; and, R-Ara-C/MTX is Rituximab 375 mg/m^2, Cytarabine 3 g/m^2 and Methotrexate 200 mg/m^2.
Arm/Group | Arm A 1mcg/kg | ARM A 3mcg/kg | Arm A 10mcg/kg | Arm B 1mcg/kg | Arm B 3mcg/kg | Arm B 10mcg/kg | Placebo
Number analyzed (Participants) | 4 | 4 | 12 | 4 | 4 | 4 | 12
K/μL | 20.3 (3.0) | 26.3 (11.1) | 24.8 (13.0) | 22.5 (8.9) | 18.3 (6.3) | 8 (2.2) | 11.3 (1.4)

2. Primary Outcome: Days Platelets Count of < 100K/μL
Description: The optimal biologic dose was defined as the dose of AMG 531 at which the greatest proportion of patients avoided grade 4 thrombocytopenia (Platelet nadir < 25K/μL) in the absence of platelet transfusion in the blinded study cycle.
Time Frame: Prior to start of treatment and then at least 2 times a week during treatment until end of cycle 2 (1 cycle = 21 days)
Measure: Mean (Standard Error); unit: days
Groups:
- Arm A 10mcg/kg: Cycle 1, Chemotherapy (R-HyperCVAD) alone.
  Cycle 2, Chemotherapy (R-Ara-C/MTX), followed by either 1 mcg/kg or 3 mcg/kg or 10 mcg/kg AMG531 subcutaneously on days -5 and 5 (Arm A)
  R-HyperCVAD alternating with R-Ara-C/MTX where R-HyperCVAD is Rituximab 375 mg/m^2; plus Cyclophosphamide 300 mg/m^2, Vincristine 1.4 mg/m^2, Doxorubicin (Adriamycin) 50 mg/m^2, and Dexamethasone 40 mg (CVAD), Mesna 600mg/m^2; and, R-Ara-C/MTX is Rituximab 375 mg/m^2, Cytarabine 3 g/m^2 and Methotrexate 200 mg/m^2.
Arm/Group | Arm A 1mcg/kg | Arm A 3mcg/kg | Arm A 10mcg/kg | Arm B 1mcg/kg | Arm B 3mcg/kg | Arm B 10mcg/kg | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 12
days | 5.5 (0.9) | 5.3 (1.1) | 8.3 (2.3) | 6.8 (1.7) | 8 (0.8) | 9.3 (2.0) | 9.8 (0.7)

ADVERSE EVENTS:
Time Frame: Toxicity assessments with each dose level/cycle (3 week cycle) up to 6 cycles; overall study treatment period four years and three months.
Arm/Group | 1 mcg/ kg AMG531 Pre & Post Chemotherapy | 3 mcg/ kg AMG531 Pre & Post Chemotherapy | 10 mcg/ kg AMG531 Pre & Post Chemotherapy | Placebo (Arm A & Arm B) With Chemotherapy | 1 mcg/ kg AMG531 Post Chemotherapy | 3 mcg/ kg AMG531 Post Chemotherapy | 10 mcg/ kg AMG531 Post Chemotherapy
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/4 | 0/14 | 0/5 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/6 | 4/4 | 4/4 | 6/14 | 1/5 | 2/4 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mcg/ kg AMG531 Pre & Post Chemotherapy (N=6) | 3 mcg/ kg AMG531 Pre & Post Chemotherapy (N=4) | 10 mcg/ kg AMG531 Pre & Post Chemotherapy (N=4) | Placebo (Arm A & Arm B) With Chemotherapy (N=14) | 1 mcg/ kg AMG531 Post Chemotherapy (N=5) | 3 mcg/ kg AMG531 Post Chemotherapy (N=4) | 10 mcg/ kg AMG531 Post Chemotherapy (N=4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 4 (4) | 4 (4) | 1 (1) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No